CLINICAL TRIAL: NCT06681883
Title: Effectiveness of a Nursing Care Program Based on the Care Bag Theory for Healthy Internet Use in Adolescents: An Action Research Study
Brief Title: Implementation of the Care Bag Theory for Healthy Internet Use in Adolescents (CHIA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Arif Özparlak, PhD, Research Assistant, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAEK-152
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Internet Addiction; Problematic Internet Use; Healthy Internet Use
Keywords: adolescent; problematic internet use; nursing; model; healthy internet use
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Action group (Experimental)
  Interventions: Behavioral: A nursing care program based on the Care Bag Theory for Healthy Internet Use in Adolescents (CHIA)

INTERVENTIONS:
Behavioral: A nursing care program based on the Care Bag Theory for Healthy Internet Use in Adolescents (CHIA) — A nursing care program based on the Care Bag Theory for Healthy Internet Use in Adolescents (CHIA)
  The nursing care program based on the CHIA model is designed for adolescents with problematic internet use. The program is grounded in the concepts of the draft model. It consists of eight sessions, each expected to last 40-50 minutes. One session will be held per week. The first session includes introductions and an overview of the program, the second session aims to strengthen the adolescent's motivation for change, the third session focuses on improving the adolescent's self-control skills, the fourth session aims to enhance family functionality, the fifth session helps develop offline activities to replace internet use, the sixth and seventh sessions work on developing coping skills, and the eighth session includes the evaluation and termination of the program.

SUMMARY:
The study aimed to investigate the effect of a nursing care program based on the Care Bag Theory for Healthy Internet Use in Adolescents (CHIA) on adolescents' problematic internet use, self-regulation, family relationships, and coping skills.

DETAILED DESCRIPTION:
This study constitutes a part of the doctoral thesis titled "Development of a Nursing Intervention Model Specific to Problematic Internet Use in Adolescents"

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreeing to participate in the study,
* Being between the ages of 12-18,
* Receiving outpatient follow-up at the Child and Adolescent Mental Health Clinic,
* Having a Problematic Internet Use (PIU) issue (PIU is assessed according to the criteria by the doctors at the clinic. The doctors refer adolescents who meet the criteria. These criteria are as follows: a) using the internet for longer than planned, b) experiencing withdrawal symptoms when unable to access the internet, c) failing to control internet usage, d) being excessively preoccupied with the internet, e) losing interest in offline hobbies, f) a desire to use the internet more, g) continuing excessive internet use despite knowing it negatively affects their life, h) using the internet to escape problems, i) lying about internet use).

Exclusion Criteria:

* Having a speech, hearing, or self-expression impairment,
* Having received or currently receiving professional support related to PIU.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Problematic Internet Use Scale-Adolescent (PIUS-A) | Data will be collected two times: pre-intervention and immediately post-intervention.
  The scale consists of 27 items and is of a five-point Likert type. The lowest possible score on the scale is 27, and the highest score is 135. Higher scores on the scale indicate that adolescents' problematic internet use has increased and become unhealthy. The PIUS-A scale has three subscales: negative consequences of internet use, excessive use, and social benefit/social comfort.

SECONDARY OUTCOMES:
The Adolescent Self Regulatory Inventory (ASRI) | Data will be collected two times: pre-intervention and immediately post-intervention.
  The scale consists of 32 items and has two subscales: 'self-control success' and 'self-control failure.' The self-control success subscale contains 18 items, while the self-control failure subscale contains 14 items. The scale uses a four-point Likert-type rating. The scale is used to calculate the total score. The lowest possible score on the ASRI is 32, and the highest score is 128. A higher score on the scale indicates that the adolescent's self-control skills are good.
Kidcope | Data will be collected two times: pre-intervention and immediately post-intervention.
  The scale consists of 11 items. The Kidcope has three subscales: Active Coping (Items 3, 6, 8, 10), Negative Coping (Items 4, 5, 7), and Avoidant Coping (Items 1, 2, 9, 11). Each subscale score is obtained by summing the relevant items in order. The possible scores range from 0 to 12 for both the Active Coping and Avoidant Coping subscales, and from 0 to 9 for the Negative Coping subscale. As the score increases, it indicates a higher use of the corresponding coping strategy.
The Family Relationship Scale for Children | Data will be collected two times: pre-intervention and immediately post-intervention.
  The scale consists of 20 items and was developed to measure how children perceive their relationships with their families. Participants respond to each item with "never" (1), "sometimes" (2), or "always" (3). The scale has two subscales: Restrictive Family Relationships and Supportive Family Relationships. Items 2, 3, 4, 5, 6, 10, 14, 16, 18, and 19 form the Restrictive Family Relationships subscale. A higher score in this subscale indicates that the child perceives the relationships within the family as restrictive. Items 1, 7, 8, 9, 11, 12, 13, 15, 17, and 20 form the Supportive Family Relationships subscale. A higher score in this subscale indicates that the child perceives the relationships within the family as supportive.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Kepez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang W, Ye J, Zhu Y, Huang D, Zhao X. Longitudinal relationship between internet self-control and problematic internet use among Chinese adolescents: mediating role of meaning in life. Front Psychiatry. 2023 Dec 7;14:1258673. doi: 10.3389/fpsyt.2023.1258673. eCollection 2023. PMID 38144476
- [Result] Shek DT, Yu L, Leung H, Wu FK, Law MY. Development, implementation, and evaluation of a multi-addiction prevention program for primary school students in Hong Kong: the B.E.S.T. Teen Program. Asian J Gambl Issues Public Health. 2016;6(1):5. doi: 10.1186/s40405-016-0014-z. Epub 2016 Jul 8. PMID 27630812
- [Result] Peterson SJ. Introduction to the nature of nursing knowledge. In S. J. Peterson and T. S. Bredow (Eds.), Middle range theories: Application to nursing research (3rd ed., pp. 3-41). Philadelphia: Lippincott Williams & Wilkins; 2013.
- [Result] Rakhmawati W, Kosasih CE, Widiasih R, Suryani S, Arifin H. Internet Addiction Among Male Adolescents in Indonesia: A Qualitative Study. Am J Mens Health. 2021 May-Jun;15(3):15579883211029459. doi: 10.1177/15579883211029459. PMID 34189970
- [Result] Paulus FW, Ohmann S, von Gontard A, Popow C. Internet gaming disorder in children and adolescents: a systematic review. Dev Med Child Neurol. 2018 Jul;60(7):645-659. doi: 10.1111/dmcn.13754. Epub 2018 Apr 6. PMID 29633243
- [Result] Park E, Kwon M. Health-Related Internet Use by Children and Adolescents: Systematic Review. J Med Internet Res. 2018 Apr 3;20(4):e120. doi: 10.2196/jmir.7731. PMID 29615385
- [Result] Ozparlak A, Karakaya D, Onder A, Gunbayi I. Problematic internet use in adolescents: A phenomenological study. J Psychiatr Ment Health Nurs. 2023 Aug;30(4):731-742. doi: 10.1111/jpm.12900. Epub 2023 Jan 31. PMID 36662598
- [Result] Marchant A, Hawton K, Stewart A, Montgomery P, Singaravelu V, Lloyd K, Purdy N, Daine K, John A. A systematic review of the relationship between internet use, self-harm and suicidal behaviour in young people: The good, the bad and the unknown. PLoS One. 2017 Aug 16;12(8):e0181722. doi: 10.1371/journal.pone.0181722. eCollection 2017. PMID 28813437
- [Result] Lyons J. Reflective education for professional practice: discovering knowledge from experience. Nurse Educ Today. 1999 Jan;19(1):29-34. doi: 10.1054/nedt.1999.0607. PMID 10222968
- [Result] Lukavska K, Hrabec O, Lukavsky J, Demetrovics Z, Kiraly O. The associations of adolescent problematic internet use with parenting: A meta-analysis. Addict Behav. 2022 Dec;135:107423. doi: 10.1016/j.addbeh.2022.107423. Epub 2022 Jul 6. PMID 35933287